CLINICAL TRIAL: NCT04462185
Title: A Prospective Cohort Study of Chinese Patients With Pulmonary Nodules: Prediction of Lung Cancer Using Noninvasive Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AnchorDx Medical Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); Shanghai Zhongshan Hospital (Other); West China Hospital (Other); Beijing Chao Yang Hospital (Other); Johnson & Johnson (China) Investment Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AnchorDx LC023
Record Dates: First submitted 2020-07-05; First posted 2020-07-08 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Nodules
Keywords: Noninvasive Biomarkers; Lung Cancer; Computed Tomography (CT); Nasal epithelium
MeSH Terms: conditions — Multiple Pulmonary Nodules; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood; Nasal epithelium; Biopsy / surgical specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: This is a prospectively enrolling cohort study and 3000 patients (1500 GGO and 1500 solid / semi solid nodules) with radiologic diagnosis of indeterminate pulmonary nodule (5-30 mm) will be recruited. All participants will be followed up with chest CT or low-dose computed tomography (LDCT) scans for 2-3 years, and take the diagnostic test, a genomic and transcriptomic landscape analysis, at each visit.
  Interventions: Diagnostic Test: A genomic and transcriptomic landscape analysis

INTERVENTIONS:
Diagnostic Test: A genomic and transcriptomic landscape analysis — A genomic and transcriptomic landscape analysis will be developed to identify and characterize the transcriptome of benign versus malignant by using RNA sequencing, and to profile cfDNA in blood samples collected from patients with pulmonary nodules.

SUMMARY:
The broad goals of this study is to identify changes in genomic landscape during transition from stage 0 to stage 1 lung cancer.

This study intends to determine whether diagnostic biomarkers measured in minimally invasive biospecimens are able to correlate molecular, clinical and imaging features to distinguish malignant from benign pulmonary nodules. The diagnostic markers once validated can be used as broad screening tools for lung cancer.

DETAILED DESCRIPTION:
The four-year study aims to recruit 3000 patients (1500 GGO and 1500 solid / semi solid nodules) in the study based on qualifying for a lung cancer screening CT or by routine CT chest with the observation of a lung nodule between 5-30mm diameter. These patients will be followed for 2~3 years and be managed according to institutional standard of care. This may involve the Chinese Thoracic Society guideline or Fleischner criteria (either 2013 or 2017 guidelines). The clinical data, CT imaging and biospecimens will be collected during each visit. Once a patient undergoes surgery, tissue samples (FFPE) from surgery will also be collected.

The gold standard for lung cancer diagnosis will be the results of bronchoscopic biopsy of lung or lymph nodes, percutaneous biopsy of lung or other organ sites, surgical biopsy or resection, or a minimum follow-up of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older, both male and female
* Willing and able to provide a written informed consent
* Radiologic diagnosis of solid indeterminate pulmonary nodule (5-30 mm) OR semi-solid (mixed density) nodule with solid component of at least 5mm OR non-solid nodule (including pGGO); must be of appropriate size at enrollment, but nodule(s) may have been first identified within 12 months prior. Furthermore, nodule(s) < 5 mm in size may have been first identified greater than 12 months prior to enrollment though it must grow into the appropriate size range (5-30 mm) within 12 months prior to enrollment. If multiple nodules were diagnosed, choose the most representative one with the longest diameter as the target lesion; if two or more nodules are of the same largest size, choose the one with the perpendicular longest diameter
* CT scan completed within 3 months prior to enrollment
* Agree to tolerate all biospecimen collection as required by protocol
* Agree to comply with standard of care follow up visits including clinical exams, diagnostic work-ups, and imaging for 2~3 years from enrollment
* Agree to fill out Patient Lung History Questionnaire

Exclusion Criteria:

* History or previous diagnosis of primary lung cancer, metastatic lung cancer, or any other non-lung cancer within 5 years (exceptions are adequately treated squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast)
* Any receipt of cytotoxic agents within the past 6 months
* Any symptoms of lung cancer (unexplained weight loss, recent hemoptysis)
* Pregnant or lactating women
* Underwent invasive biopsy procedures (e.g. bronchoscopies or CT-guided transthoracic biopsies) before enrollment
* Receipt of transfusion within 30 days prior to enrollment
* Fail to understand or provide a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with pulmonary nodules diagnosed by chest CT or low-dose computed tomography (LDCT) scans between 5-30 mm diameter
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The changes in genomic landscape related to progression from Stage 0 to Stage I lung cancer that could be utilized for early lung cancer diagnosis and intervention. | 3 Years
  The transcriptome of benign versus malignant by using RNA sequencing. The cfDNA in blood samples collected from patients with pulmonary nodules.

SECONDARY OUTCOMES:
The biomarker changes in nasal epithelium and matching blood and tissue samples so as to validate molecular tests using nasal epithelium to predict lung cancer. | 3 Years
  The biomarker change in nasal epithelium to predict lung cancer.
The individual or combinations of clinical, molecular, and imaging features can reliably identify individuals with indeterminate lung nodules 5-30 mm who have lung cancer | 3 Years
  The individual or combination of clinical, molecular, and imaging features can reliably identify individuals who have lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan ZHONG, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (6):
- China (6):
  - Department of Respiratory and Critical Care Medicine, Beijing Chaoyang Hospital, Beijing
  - Department of Respiratory Medicine, West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Department of Respiratory, Qilu Hospital, Shandong University, Jinan
  - Department of Pulmonary Medicine, Zhongshan Hospital, Fudan University, Shanghai
  - Department of Respiratory and Critical Care Medicine, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No